CLINICAL TRIAL: NCT06757465
Title: The Effect of Counseling Grounded in Watson's Human Caring Theory on Reproductive Concerns in Women Diagnosed with Cancer: a Randomized Controlled Study
Brief Title: Women Diagnosed with Cancer & Reproductive Concerns & Watson's Human Caring Theory &Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ruken Yağız Altıntaş, Doctoral Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-1669200
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Reproductive Health
Keywords: Cancer; Counseling; Reproductive Concerns; Women
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a single-blind, randomized controlled clinical trial, parallel
Who Masked: Investigator
Masking Description: The randomization list for the study sample size of 50 women was created by a statistician. According to the list, women were divided into two groups as intervention (A) and control (B). Data were collected by a fellow who was not in the study. The fellow responsible for the data collection process collected the data without knowing which group the participants belonged to. This approach was preferred to prevent bias in the measurements and to increase the reliability of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Counseling for reproductive concerns in women diagnosed with cancer (Experimental): In this study, a total of 75 interviews were conducted with 25 participants in the intervention group in three sessions. During the interviews, counseling training based on Watson IBK developed by the researchers was applied. Each session lasted between 30-45 minutes per participant. The first session was conducted face-to-face, and the second and third sessions were conducted using online platforms within the scope of telehealth applications. Sessions were structured according to the individual needs of the participants and the durations were arranged flexibly when necessary. Immediately after the sessions of counseling training based on Watson IBC were applied, the "the Reproductive Concerns After Cancer Scale " and "the Patient Satisfaction Evaluation Form Based on Watson's Processes of Healin" were applied as interim tests to measure the effect of counseling on reproductive concerns levels of the patients. These tests were repeated 4 weeks after the end of the training.
  Interventions: Other: Counseling education based on Watson's Theory of Human Caring
- Control (No Intervention): No intervention was made to the participants in the control group after the pre-test was applied as part of the data collection process. The women in the control group received the standard counseling service routinely applied in the clinic.
  After the patients were met, detailed information about the study was given, their informed consent was obtained and the contact information of the researcher was provided to them. 4 weeks after the pre-test, "the Reproductive Concerns After Cancer Scale" and "the Patient Satisfaction Evaluation Form Based on Watson's Processes of Healing" were applied to the participants in the control group as a post-test.

INTERVENTIONS:
Other: Counseling education based on Watson's Theory of Human Caring — In this study, a total of 75 interviews were conducted with 25 participants in the intervention group in three sessions. During the interviews, counseling training based on Watson IBK developed by the researchers was applied. Each session lasted between 30-45 minutes per participant. The first session was conducted face-to-face, and the second and third sessions were conducted using online platforms (Zoom, Microsoft Teams, WhatsApp video call) within the scope of telehealth applications. Sessions were structured according to the individual needs of the participants and the durations were arranged flexibly when necessary. Telehealth applications provided easy access to the participants during the counseling process and supported the continuity of individual counseling services.
  Arms: Counseling for reproductive concerns in women diagnosed with cancer

SUMMARY:
This is a single-blind randomized controlled experimental study with a pre-test post-test design to examine the effects of counseling based on Watson's Human Caring Theory given to women between the ages of 18-45 diagnosed with cancer on fertility concerns.

DETAILED DESCRIPTION:
Reproductive concerns, one of the important problems affecting the quality of life of women diagnosed with cancer, is becoming a critical problem that needs to be addressed with both psychological and social dimensions when combined with concerns about the future. This study aims to examine the effect of counseling on reproductive concerns in women diagnosed with cancer, based on Watson's Human Caring Theory and an interview guide prepared by the researcher.

A randomized controlled experimental study with a pre-test-post-test design was conducted to examine the effects of counseling based on Watson's Human Caring Theory given to women between the ages of 18-45 diagnosed with cancer on reproductive concerns. The universe of the study consisted of female patients diagnosed with cancer between the ages of 18-45 who applied to the Department of Obstetrics and Gynecology (Family Planning and Infertility Research and Application Center and Gynecology Oncology Clinic), Oncology Department and General Surgery Department of Ege University Hospital. The research was conducted in the designated clinics of Ege University Faculty of Medicine Hospital between January 1, 2024 and September 15, 2024. The sample of the research consisted of 50 women diagnosed with cancer, 25 intervention and 25 controls. In the data collection process of the study, a "Participant Information Form" and a " "Reproductive Concerns After Cancer Scale" will be administered in the pre-test for both intervention and control groups. For the control group, four weeks after the pre-test, the "Reproductive Concerns After Cancer Scale" and the "Patient Satisfaction Evaluation Form According to Watson's Healing Processes" will be applied. For the intervention group, counseling sessions grounded in Watson's Human Caring Theory will be conducted in three sessions, and a post-test will be administered four weeks later.

The study, it was determined that the reproductive concerns levels of women in the intervention group who received counseling education based on Watson's Theory of Human Caring were significantly lower (p < 0.05). The patient satisfaction assessment scores based on the improvement processes showed a statistically significant difference between the intervention and control groups. The scores of the intervention group were found to be higher compared to the control group (p < 0.05). The Patient Satisfaction Evaluation Form scores based on Watson's Processes of Healing showed a statistically significant difference between the intervention and control groups. The scores of the intervention group were found to be higher compared to the control group (p < 0.05). Counseling based on Watson's Theory of Human Caring was found to reduce reproductive concerns and improve patient satisfaction based on Watson's Processes of Healing in women diagnosed with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being of reproductive age between 18-45 years,
* Not starting chemotherapy and radiotherapy treatment,
* Having no vision, hearing or mental problems,
* Knowing how to read and write and speaking Turkish,
* Agreeing to participate in the study voluntarily.

Exclusion Criteria:

* Being in menopause,
* Having had a hysterectomy,
* Being in Stage IV of the cancer diagnosed.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
The Reproductive Concerns After Cancer Scale | Change from before implementation and 4th week of practice.
  The scale assesses fertility and parenting concerns. It consists of 18 items. The lowest total score from the scale is 18 and the highest is 90. As the score increases, the level of reproductive concerns increases.
The Patient Satisfaction Evaluation Form Based on Watson's Processes of Healing | Change from 4th week of practice.
  It is used to evaluate nursing care based on Watson's Human Caring Theory. It consists of 6 questions. The total highest score from this evaluation form is 35, and the lowest score is five.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to publish it as an article.
Supporting Information: Study Protocol
Time Frame: from July 2025
Access Criteria: It is planned to be published in an open access journal.

REFERENCES:
- [Background] Qiu J, Tang L, Li P, Fu J. An investigation into the reproductive concerns of young women with breast cancer. Asia Pac J Oncol Nurs. 2022 Mar 24;9(6):100055. doi: 10.1016/j.apjon.2022.03.007. eCollection 2022 Jun. PMID 35615663
- [Background] Xiao Y, Li J, Lei J, Li X, Hu M, Zhao J, Han L, Chen O. Qualitative study of the fertility information support experiences of young breast cancer patients. Eur J Oncol Nurs. 2023 Feb;62:102275. doi: 10.1016/j.ejon.2023.102275. Epub 2023 Jan 25. PMID 36716530
- [Background] Young K, Shliakhtsitsava K, Natarajan L, Myers E, Dietz AC, Gorman JR, Martinez ME, Whitcomb BW, Su HI. Fertility counseling before cancer treatment and subsequent reproductive concerns among female adolescent and young adult cancer survivors. Cancer. 2019 Mar 15;125(6):980-989. doi: 10.1002/cncr.31862. Epub 2018 Nov 29. PMID 30489638